CLINICAL TRIAL: NCT07253259
Title: A Clinical Study Evaluating the Safety and Efficacy of GT729 Universal Cell Injection in the Treatment of Refractory or Relapsed Chronic Graft-versus-host Disease (cGVHD)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Collaborators: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CD-CHN-729-001
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: cGVHD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GT729 Injection treatment group (Experimental): GT729 Injection
  Interventions: Biological: GT729 Injection

INTERVENTIONS:
Biological: GT729 Injection — GT729 Injection

SUMMARY:
The goal of this clinical study is to evaluate the safety and efficacy of GT729 universal cell injection in the treatment of refractory or relapsed chronic graft-versus-host disease (cGVHD).

ELIGIBILITY:
Inclusion Criteria:

* Participants or their legal representatives voluntarily sign a written informed consent form, are willing and able to comply with the procedures of this study.
* Aged 18 to 65 years old (inclusive) when signing the informed consent, regardless of gender.
* Participants must meet the following criteria:

  1. The subjects are allogeneic hematopoietic stem cell transplantation (alloHSCT) recipients with active chronic graft-versus-host disease (active cGVHD) requiring systemic immunosuppressive therapy.
  2. The subjects are patients with refractory or relapsed active cGVHD after receiving at least two lines of systemic treatment.
* The laboratory test results during the screening period must meet the following criteria (except for indicators related to the study disease):

  1. Neutrophil count ≥ 1.0×10⁹/L;
  2. Hemoglobin ≥ 80g/L; Platelet count ≥ 30×10⁹/L;
  3. Alanine transaminase ≤ 3×upper limit of normal (ULN); Aspartate transaminase ≤ 3×ULN; Total bilirubin (TBIL) < 2×ULN;
  4. Creatinine clearance rate ≥ 30 mL/min.
* Women of childbearing age must:

At the time of screening, as confirmed by the investigator, the result of the serum β-human chorionic gonadotropin (β-hCG) pregnancy test is negative.

Exclusion Criteria:

* Evidence of recurrence of underlying malignant tumors or post-transplant lymphoproliferative disorder (PTLD) at the time of screening
* Having a history of severe hypersensitivity or allergies
* Suffering from the following heart diseases:

  1. New York Heart Association (NYHA) Class III or IV congestive heart failure;
  2. A myocardial infarction occurred or coronary artery bypass surgery was performed within 6 months before the screening period.
* Participants with clinically significant bleeding symptoms or a clear bleeding tendency within the 6 months prior to screening;
* Participants with severe underlying medical conditions at the time of screening;
* Participants who have undergone major surgery within 8 weeks prior to screening or are scheduled to undergo surgery during the study period;
* History of organ transplantation;
* According to the investigator's judgment, there are circumstances that would prevent the participant from completing the entire trial, confuse the trial results, or make participation in the trial not in the best interest of the participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants experiencing dose limiting toxicity | 28 days
  Proportion of participants experiencing dose limiting toxicity (DLT) within 28 days after cell infusion
Incidence of adverse events | From infusion to the end of the treatment at 24 months
  Incidence of adverse events per NCI-CTCAE version 5.0

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 6 months post infusion
  To evaluate the percentage of participants who have a confirmed partial response or complete response among total number of evaluable participants as assessed by the investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No